DIPARTIMENTO INTERAZIENDALE DI CHIRURGIA Unità Operativa di Chirurgia Generale Provinciale Direttore Prof. Carlo FEO

Ferrara, 05/11/2021

## **OFFICIAL TITLE**

The efficacy of near-infrared fluorescent cholangiography during emergency laparoscopic cholecystectomy in patients with acute cholecystitis and in difficult cholecystectomies.

## 1. BACKGROUND

Laparoscopic cholecystectomy is one of the most frequently performed surgical procedures in the Western world, with over 750,000 surgeries in the United States alone [1]. Iatrogenic bile duct injuries represent a serious and feared complication, leading to a significant increase in morbidity and mortality, healthcare costs, and medico-legal consequences [2-4]. In most cases, iatrogenic bile duct injuries are related to an altered perception of the true extrahepatic biliary anatomy, regardless of the surgeon's experience and age. Since laparoscopic cholecystectomy became the "gold standard" for treating symptomatic gallstone disease and acute cholecystitis, the incidence of iatrogenic bile duct injuries has exponentially increased. The incidence rate of major bile duct injuries ranges between 0.25% and 1%, according to the latest literature data [2-4]. The use of intraoperative cholangiography (IOC) is a way to correctly visualize the extrahepatic biliary tree (reducing the risk of iatrogenic injuries) and to identify possible associated choledocholithiasis. The routine or selective use of intraoperative cholangiography is still debated today. It is certainly true that the method has a significant morbidity rate and requires adequate equipment, which can be costly. The advent of less invasive and certainly more economical alternative methods, such as near-infrared fluorescence cholangiography (NIRF-C), could reduce costs and allow the surgery to be performed with a lower morbidity rate. Fluorescence cholangiography uses an infrared system that allows the intraoperative visualization of the extrahepatic biliary tree through the intravenous administration of a vital dye, indocyanine green (ICG). The intravenous use of this dye before laparoscopic cholecystectomy is part of routine clinical practice, and its efficacy has been confirmed in several studies in the literature [5-7]. The



correct anatomical identification of the bile ducts allows the surgeon to operate with greater safety, reducing the risk of iatrogenic injuries and the conversion rate. The method is extremely safe and poses no additional risks to the patient.

Early laparoscopic cholecystectomy also represents the "gold standard" for patients with mild (grade I) and moderate (grade II) acute cholecystitis who do not respond to initial conservative treatment if performed within 24-72 hours from symptom onset, according to the 2018 Tokyo Guidelines [8].

Fluorescence cholangiography may be challenging in an emergency setting, as inflammation and adhesions of the hepatoduodenal ligament can impair the identification of biliary structures during dissection. Achieving the so-called "critical view of safety" (CVS) can be particularly difficult in such situations.

In a recent meta-analysis, Dip F *et al.* [9] demonstrated that the use of fluorescence cholangiography during elective cholecystectomy reduces iatrogenic bile duct injuries and the conversion rate to open surgery compared to traditional white-light surgery. However, there is limited data on its feasibility and clinical impact in urgent acute cholecystitis cases. The identification of biliary structures can be challenging, especially in cases with extensive adhesions and severe inflammation, including necrosis, of the gallbladder wall and surrounding tissues.

Currently, there is little evidence regarding the effectiveness of fluorescence cholangiography during emergency laparoscopic cholecystectomies for acute cholecystitis. Only two cohort studies [10,11], an international European registry [12], and a randomized controlled trial (RCT), including elective and emergency cholecystectomies [13] have been published. In a large retrospective study involving 184 consecutive patients, Daskalaki E *et al.* [11] reported the results of 24 patients undergoing robotic cholecystectomy with ICG fluorescence for acute and gangrenous cholecystitis. The authors evaluated the percentage of visualization of four biliary structures, particularly the cystic duct (CD), common hepatic duct (CHD), common bile duct (CBD), and cystic duct-common hepatic duct junction (CD-CHD). In this subgroup of patients, the cystic duct (CD), CHD, CBD, and CD-CHD were successfully visualized in 91.6%, 79.1%, 79.1%, and 75% of cases, respectively.

Agnus V et al. [12] reported the results of the Euro-FIGS (Fluorescence-Image Guided-Surgery) European registry proposed by IRCAD center in Strasbourg in collaboration with the European Association of



Endoscopic Surgery (EAES), which enrolled 314 cases from 12 European surgical centers, including patients with symptomatic cholelithiasis (n= 248) and patients with acute cholecystitis (n= 58). A 5-point Likert scale was used to evaluate the quality of biliary anatomy visualization before and after dissection of the hepatocystic triangle during laparoscopic cholecystectomy with infrared devices. When comparing the two groups (cholelithiasis vs. acute cholecystitis), lower quality visualization scores were obtained for the CD ( $2.76 \pm 1.9$  vs.  $3.54 \pm 1.6$ , P = 0.001) and the CD-CHD junction ( $2.43 \pm 2$  vs.  $3 \pm 1.9$ , P = 0.04) before preliminary Calot dissection. The impact of inflammation on the ability to visualize the biliary tree was also confirmed through multivariate linear regression analysis.

Similar data was reported in a single-blind randomized controlled trial [13] comparing the effectiveness of fluorescence cholangiography versus white light alone. The authors demonstrated that the degree of cholecystic inflammation is the most important variable, affecting not only the visualization of CD and CBD before and after dissection, but also the visualization of the cystic-infundibulum junction after complete dissection.

The utility of NIRF-C was also confirmed by Yoshiya S *et al.* [14] during LC after percutaneous transhepatic gallbladder drainage in patients with severe acute cholecystitis. The ICG fluorescence cholangiography group showed a significantly shorter operative time, lower conversion rate, and lower rate of subtotal cholecystectomy [13].

### 2. SIGNIFICANCE OF THE STUDY

This is a prospective observational cohort study of patients who underwent emergency laparoscopic cholecystectomy for acute cholecystitis. The study aims to to evaluate the efficacy of NIRF-C for real-time visualization of the biliary tree in emergency laparoscopic cholecystectomy at a regional health care center (Delta Hospital, AUSL of Ferrara, University of Ferrara, Italy) before and after hepatocystic triangle dissection and in different degrees of severity of acute cholecystitis according to the American Association of Surgery for Trauma (AAST) classification, specifically distinguishing between non-gangrenous (grade I) and gangrenous or complicated (grades II-V) forms.

## 2. STUDY POPULATION. INCLUSION AND EXCLUSION CRITERIA.

The study population consist of patients with lithiasic and alithiasic acute cholecystitis.



**Inclusion criteria:** a) Patients aged >18 years-old with a clinical and ultrasound diagnosis of acute cholecystitis who underwent laparoscopic cholecystectomy within 24-72 hours from symptom onset. b) Operable patients (ASA score 0-3).

**Exclusion criteria:** a) Patients with known allergy to indocyanine green. b) ASA score 4-5. c) Patients not operable with a laparoscopic approach due to high cardiopulmonary risk. d) Previous biliary tract surgeries. e) History of liver cirrhosis or severe liver disease. f) Pregnant and/or breastfeeding patients.

## 3. STUDY DESIGN AND DESCRIPTION

## **Primary objectives:**

Rate of correct visualization of extrahepatic bile ducts (CD, CHD, CBD, CD, CHD junction, and any
accessory or aberrant ducts) in different severity degrees of acute cholecystitis according to the
AAST classification, particularly distinguishing non-gangrenous forms (grade I) from gangrenous
and complicated forms (grades II-V).

# **Secondary objectives:**

- Conversion rate;
- Bail-out procedures (such as subtotal cholecystectomy, antegrade cholecystectomy);
- Iatrogenic bile duct injuries;
- Total surgery duration;
- Post-operative complications rate (30 days);
- Length of hospital stay;
- 30-day mortality.

The study will involve the systematic use of fluorescence cholangiography during all laparoscopic cholecystectomy procedures for acute cholecystitis, with the intravenous administration of the vital dye



Verdye 45-60 minutes before surgery at a dosage of 0.05 mg/kg or 2.5 mg/dL, according to the recent guidelines of the International Society for Fluorescence Guided-Surgery (ISFGS) and the latest consensus conference published in Annals of Surgery 2021 [16]. The patient will sign an informed consent form regarding the administration of the vital dye, with all relevant information about the method, possible benefits, and risks. The patient will also have the option to withdraw from the study at any time without affecting the care they receive. The equipment used will be Stryker's fluorescence imaging system (Stryker, Portage, Miami, USA): the systems has a 10-mm laparoscope, a camera head, a xenonlight guide cable, a video processor/illuminator, and a high-definition monitor. The charge-coupled device camera and the xenon light source could filter out light with wavelengths below 810 nm and above 800 mm. The laparoscope was able to transmit near-infrared light, allowing images to be switched from full color to fluorescence images. At the end of each procedure, the operator will fill out a form reporting the following data:

a) Patient's demographic data (surname, name, age, gender); b) B.M.I. (Body Mass Index); c) Previous cholangio-MR and/or ERCP; d) Surgeon's experience (defined as more than 50 laparoscopic cholecystectomy procedures performed); e) Biliary structures visualized after administration of the vital dye before and after dissection of Calot's triangle; f) Identification of any biliary anomalies, accessory or aberrant ducts; g) Time taken to achieve CVS; h) Total surgery duration; i) Possible conversion to open surgery; j) Any minor and/or major complications; k) Need for and use of any additional drains; l) Total length of postoperative hospital stay; m) 30-day mortality.

The study data will be collected by authorized personnel and analyzed in compliance with the current European privacy regulations, safeguarding patient confidentiality. The study will be performed in accordance with the Declaration of Helsinki guidelines.

## 4. STATISTICAL ANALYSIS

All collected data will be included in a study-specific database and analyzed using MedCalc 20.011 (Ostend, Belgium). Descriptive statistics were used to characterize the population, including proportions, medians, means  $\pm$  standard deviations (SDs), and ranges. The two-tailed Chi-square test was used for the statistical comparison of proportions. The Chi-square test was used to compare the proportion of successful FC visualization (i.e., visualization rates) of the biliary tree (cystic duct [CD], common hepatic duct [CHD], and common bile duct [CBD]) before and after Calot's dissection in all patients. Comparisons of the proportion



of successful FC visualization of the biliary tree were performed by comparing the different degrees of acute cholecystitis according to the intra-operative AAST classification. A P-value <0.05 was considered statistically significant.

# **5. STUDY DURATION**

The study will last 18-24 months.

## 6. FINANCIAL ASPECTS

The study is not for profit and is carried out without external funding.

## 7. INSURANCE

No specific insurance is required.

### 8. APPROVAL OF THE LOCAL ETHICS COMMITTEE

The study will be conducted in accordance with the Declaration of Helsinki, the European Union Medical Device Directive (93/42/ECC art.15), and the local transpositions of the Member States. The study will be carried out in accordance with the guidelines for clinical studies as outlined in EN ISO 14155 and in compliance with good clinical practice. It will start after obtaining the favorable opinion of the local Ethics Committee.

# 9. RESPONSIBLE FOR DATA MANAGEMENT AND METHODS OF DATA EVALUATION AND PROCESSING

The study Principal Investigator (P.I.) is Prof. Carlo Vittorio Feo; the data management will be overseen by Dr. Antonio Pesce, as co-principal investigator and study director.

### **REFERENCES**

- Way LW, Stewart L, Gantert W, Liu K, Lee CM, Whang K, Hunter JG. Causes and prevention of laparoscopic bile duct injuries: analysis of 252 cases from a human factors and cognitive psychology perspective. *Ann Surg* 2003; 237: 460-469 [PMID: 12677139 DOI: 10.1097/01.SLA.0000060680.92690.E9]
- **2. Nuzzo G**, Giuliante F, Giovannini I, Ardito F, D'Acapito F, Vellone M, Murazio M, Capelli G. Bile duct injury during laparoscopic cholecystectomy: results of an Italian national survey on 56 591 cholecystectomies. *Arch Surg* 2005; **140**: 986-992 [PMID: 16230550 DOI: 10.1001/archsurg.140.10.986]
- **3. Pesce A**, Portale TR, Minutolo V, Scilletta R, Li Destri G, Puleo S. Bile duct injury during laparoscopic cholecystectomy without intraoperative cholangiography: a retrospective study on 1,100 selected patients. *Dig Surg* 2012; **29**: 310-314 [PMID: 22986956 DOI: 10.1159/000341660]
- **4. Pesce A**, Palmucci S, La Greca G, Puleo S. Iatrogenic bile duct injury: impact and management challenges. *Clin Exp Gastroenterol* 2019; **12**: 121-128 [PMID: 30881079 DOI: 10.2147/CEG.S169492]
- **5. Pesce A**, Latteri S, Barchitta M, Portale TR, Di Stefano B, Agodi A, Russello D, Puleo S, La Greca G. Near-infrared fluorescent cholangiography real-time visualization of the biliary tree during elective laparoscopic cholecystectomy. HPB (Oxford). 2018 Jun;20(6):538-545.
- **6. Pesce A**, Piccolo G, La Greca G, Puleo S. Utility of fluorescent cholangiography during laparoscopic cholecystectomy: A systematic review. *World J Gastroenterol* 2015; **21**: 7877-7883 [PMID: 26167088 DOI: 10.3748/wjg.v21.i25.7877]
- **7. Pesce A**, Piccolo G, Lecchi F, Fabbri N, Diana M, Feo CV. Fluorescent cholangiography: An up-to-date overview twelve years after the first clinical application. *World J Gastroenterol* 2021; 27(36): 5989-6003 [DOI: 10.3748/wjg.v27.i36.5989]
- **8. Okamoto K**, Suzuki K, Takada T, Strasberg SM, Asbun HJ, Endo I, Iwashita Y, Hibi T, Pitt HA, Umezawa A, Asai K, Han HS, Hwang TL, Mori Y, Yoon YS, Huang WS, Belli G, Dervenis C, Yokoe M, Kiriyama S, Itoi T, Jagannath P, Garden OJ, Miura F, Nakamura M, Horiguchi A, Wakabayashi G, Cherqui D, de Santibañes E, Shikata S, Noguchi Y, Ukai T, Higuchi R, Wada K, Honda G, Supe AN, Yoshida M, Mayumi T, Gouma DJ, Deziel DJ, Liau KH, Chen MF, Shibao K, Liu KH, Su CH, Chan ACW, Yoon DS, Choi IS, Jonas E, Chen XP, Fan ST, Ker CG, Giménez ME, Kitano S, Inomata M, Hirata K, Inui K, Sumiyama Y, Yamamoto M. Tokyo Guidelines 2018:

flowchart for the management of acute cholecystitis. *J Hepatobiliary Pancreat Sci* 2018; **25**: 55-72 [PMID: 29045062 DOI: 10.1002/jhbp.516]

- **9. Dip F**, Lo Menzo E, White KP, Rosenthal RJ. Does near-infrared fluorescent cholangiography with indocyanine green reduce bile duct injuries and conversions to open surgery during laparoscopic or robotic cholecystectomy? *Surgery* 2021; **169**: 859-867 [PMID: 33478756 DOI:10.1016/j.surg.2020.12.008]
- **10. Di Maggio F**, Hossain N, De Zanna A, Husain D, Bonomo L. Near-Infrared Fluorescence Cholangiography can be a Useful Adjunct during Emergency Cholecystectomies. *Surg Innov* 2020; 1553350620958562 [PMID: 32936054 DOI: 10.1177/1553350620958562]
- **11. Daskalaki D**, Fernandes E, Wang X, Bianco FM, Elli EF, Ayloo S, Masrur M, Milone L, Giulianotti PC. Indocyanine green (ICG) fluorescent cholangiography during robotic cholecystectomy: results of 184 consecutive cases in a single institution. *Surg Innov* 2014; **21**: 615-621 [PMID: 24616013 DOI: 10.1177/1553350614524839]
- **12. Agnus** V, Pesce A, Boni L, Van Den Bos J, Morales-Conde S, Paganini AM, Quaresima S, Balla A, La Greca G, Plaudis H, Moretto G, Castagnola M, Santi C, Casali L, Tartamella L, Saadi A, Picchetto A, Arezzo A, Marescaux J, Diana M. Fluorescence-based cholangiography: preliminary results from the IHU-IRCAD-EAES EURO-FIGS registry. *Surg Endosc* 2020; **34**: 3888-3896 [PMID: 31591654 DOI: 10.1007/s00464-019-07157-3]
- **13. Dip F**, LoMenzo E, Sarotto L, Phillips E, Todeschini H, Nahmod M, Alle L, Schneider S, Kaja L, Boni L, Ferraina P, Carus T, Kokudo N, Ishizawa T, Walsh M, Simpfendorfer C, Mayank R, White K, Rosenthal RJ. Randomized Trial of Near-infrared Incisionless Fluorescent Cholangiography. *AnnSurg* 2019; **270**: 992-999 [PMID: 30614881 DOI: 10.1097/SLA.0000000000003178]
- **14. Yoshiya S**, Minagawa R, Kamo K, Kasai M, Taketani K, Yukaya T, Kimura Y, Koga T, Kai M, Kajiyama K, Yoshizumi T. Usability of Intraoperative Fluorescence Imaging with Indocyanine Green During Laparoscopic Cholecystectomy After Percutaneous Transhepatic Gallbladder Drainage. *WorldJ Surg* 2019; **43**: 127-133 [PMID: 30105635 DOI: 10.1007/s00268-018-4760-1]
- **15. Strasberg SM**, Hertl M, Soper NJ. An analysis of the problem of biliary injury during laparoscopic cholecystectomy. J Am Coll Surg. 1995 Jan;180(1):101-25. PMID: 8000648.
- **16. Wang X**, Teh CSC, Ishizawa T, Aoki T, Cavallucci D, Lee SY, Panganiban KM, Perini MV, Shah SR, Wang H, Xu Y, Suh KS, Kokudo N. Consensus Guidelines for the Use of Fluorescence Imaging in Hepatobiliary Surgery. Ann Surg. 2021 Jul 1;274(1):97-106. doi: 10.1097/SLA.0000000000004718. PMID: 33351457.

Vace

Prof. Carlo FEO

UOC di Chirurgia Generale Provinciale, Azienda USL di Ferrara,

Via Valle Oppio, 2, Lagosanto, Ferrara

Dipartimento di Scienze mediche - Università degli Studi di Ferrara

Email: fcl@unife.it

Dr Antonio PESCE

UOC di Chirurgia Generale Provinciale, Azienda USL di Ferrara,

Via Valle Oppio, 2, Lagosanto, Ferrara

Dipartimento di Scienze mediche - Università degli Studi di Ferrara

Email: antonio.pesce@unife.it



#### Comitato Etico di Area Vasta Emilia Centro

Il Comitato Etico di Area Vasta Emilia Centro della Regione Emilia-Romagna (CE-AVEC) è stato istituito presso IRCCS Azienda Ospedaliero-Universitaria di Bologna, Policlinico S.Orsola-Malpighi con delibera n. 6 del 10/1/2018. Il CE-AVEC opera in conformità al DM 12/05/2006 e al DM 08/02/2013.

Bologna, 16/12/2021

# 1034/2021/Oss/AUSLFe valutato nella seduta del 16/12/2021

Prof. Carlo Feo Direttore U.O. Chirurgia Generale Provinciale Ospedale del Delta AUSL Ferrara cvfeo@unife.it

Oggetto: L'efficacia della colangiografia fluorescente (NIRF-C) durante colecistectomia videolaparoscopica in urgenza nei pazienti affetti da colecistite acuta e nelle colecistectomie difficili

Codice Protocollo: Colecistiti Acute

Codice interno CE: 1034/2021/Oss/AUSLFe

Promotore: Azienda USL di Ferrara Centro Coordinatore: monocentrico

Sperimentatore Responsabile: Prof. Carlo Feo

Centro clinico: U.O. Chirurgia Generale Provinciale, Ospedale del Delta - Azienda USL di

Ferrara

## Elenco della documentazione esaminata:

Lettera di Trasmissione

Protocollo di studio

Sinossi dello studio

Foglio informativo

Consenso allo studio

Consenso al trattamento dati

CRF scheda raccolta dati

CV dello sperimentatore locale aggiornato e firmato (Prof. Carlo Feo)

Dichiarazione di assenza di conflitto di interesse

Modulo di fattibilità

Allegato: elenco dei componenti del Comitato Etico presenti al momento dell'espressione del presente parere

**NOTA:** per qualsiasi successiva comunicazione relativa allo studio in oggetto è indispensabile fare riferimento al codice interno CE che identifica lo studio (indicato nell'oggetto) e alla data della seduta di valutazione.



Comitato Etico di Area Vasta Emilia Centro

Il Comitato Etico di Area Vasta Emilia Centro della Regione Emilia-Romagna (CE-AVEC) è stato istituito presso IRCCS Azienda Ospedaliero–Universitaria di Bologna, Policlinico S.Orsola-Malpighi con delibera n. 6 del 10/1/2018. Il CE-AVEC opera in conformità al DM 12/05/2006 e al DM 08/02/2013.

Il Comitato Etico, nella seduta telematica del giorno 16/12/2021, esprime all'unanimità parere favorevole alla conduzione dello studio a condizione che sia dato riscontro alle sottoriportate richieste.

Relativamente all'informativa per la partecipazione allo studio (vedi allegato):

- la parte evidenziata in giallo usa termini troppo tecnici e sembra copiata dal protocollo. Occorre semplificare e sintetizzare, indicando inoltre semplicemente il numero dei soggetti partecipanti;
- deve essere descritto cosa avverrà durante la procedura oggetto di studio, specificando che si tratta di procedura routinaria (se così è);
- deve essere spiegato al/alla paziente che, rispetto alla pratica clinica standard, l'unica differenza è che verranno raccolti in modo sistematico una serie di dati che riguardano lui/lei e la procedura.

Si reputa opportuno produrre e presentare anche la lettera per il medico di medicina generale.

La documentazione sopra indicata (contrassegnata, ove applicabile, da una nuova versione e fornita anche in versione con revisioni in evidenza) dovrà essere inviata al Comitato Etico che ne verificherà la correttezza. Resta inteso che l'avvio dello studio è subordinato alla ricezione di quanto sopra.

Si precisa che

- Lo studio potrà essere avviato solo dopo aver ricevuto il nulla osta da parte della Direzione Generale della struttura sanitaria di riferimento ai sensi dell'art. 7 della L.R. n. 9/2017;
- ai fini del monitoraggio dell'andamento dello studio in oggetto, lo Sperimentatore Responsabile dovrà comunicare al Comitato Etico le seguenti informazioni relativamente a questo singolo centro sperimentale: data di inizio arruolamento, data di fine arruolamento e data di conclusione dello studio. In ogni caso, a partire dall'anno di approvazione dello studio e fino alla sua conclusione, almeno una volta all'anno e comunque entro e non oltre il 31 dicembre, dovrà essere fornito un rapporto annuale sullo stato di avanzamento dello studio. Per le suddette comunicazioni è possibile utilizzare il modulo disponibile sul sito web del Comitato Etico (https://www.aosp.bo.it/files/modulo monitoraggio ceavec v3 5-7-19 def.doc). Il modulo compilato, firmato e datato, andrà inviato esclusivamente in formato elettronico all'indirizzo email dedicato monitoraggiostudi@ospfe.it indicando nell'oggetto il nome dello Sperimentatore Responsabile locale ed il codice assegnato dal Comitato allo studio.

Cordiali saluti

IL PRESIDENTE

Allegato: elenco dei componenti del Comitato Etico presenti al momento dell'espressione del presente parere

**NOTA:** per qualsiasi successiva comunicazione relativa allo studio in oggetto è indispensabile fare riferimento al codice interno CE che identifica lo studio (indicato nell'oggetto) e alla data della seduta di valutazione.



### Comitato Etico di Area Vasta Emilia Centro

Il Comitato Etico di Area Vasta Emilia Centro della Regione Emilia-Romagna (CE-AVEC) è stato istituito presso IRCCS Azienda Ospedaliero-Universitaria di Bologna, Policlinico S.Orsola-Malpighi con delibera n. 6 del 10/1/2018. Il CE-AVEC opera in conformità al DM 12/05/2006 e al DM 08/02/2013.

### Componenti Comitato Etico Area Vasta Emilia Centro (CE-AVEC) Seduta telematica del 16/12/2021

| Nome e Cognome | Qualifica secondo il DM 8/02/2013 | Struttura di<br>appartenenza | Presente/<br>Assente |
|---|---|---|---|
| Primiano Iannone * -<br>Presidente | Clinico specialista in medicina interna/gastroenterologia | Istituto Superiore di Sanità | P |
| Elisabetta Poluzzi -<br>Vicepresidente | Farmacologo | Università degli Studi di<br>Bologna | P |
| Lucia Alberghini | Farmacista del Servizio Sanitario<br>Regionale | AUSL di Bologna | Р |
| Federica Banorri | Esperto in materia giuridica | IRCCS AOU di Bologna | A |
| Gianluca Calogero Campo | Cardiologo, esperto di nuove procedure tecniche, diagnostiche e terapeutiche, invasive e semi invasive | AOU di Ferrara/Università<br>degli Studi di Ferrara | Р |
| Edoardo Carretto * | Clinico specialista in malattie infettive e microbiologia | AUSL di Reggio Emilia<br>IRCCS | P |
| Fausto Catena * | Clinico specialista in chirurgia | AUSL della Romagna | P |
| Alessandra Cerioli * | Rappresentante del volontariato o dell'associazionismo di tutela dei pazienti | Lega Italiana per la lotta<br>contro l'AIDS (LILA) | Р |
| Paolo Cristiani * | Clinico specialista in ginecologia | Libero professionista | Р |
| Viola Damen | Direttore Sanitario dell'Istituto<br>Ortopedico Rizzoli | Istituto Ortopedico Rizzoli di<br>Bologna | Α |
| Piero De Carolis | Clinico specialista in neurologia | Libero professionista | P |
| Alessandra De Palma | Medico legale | IRCCS AOU di Bologna | Р |
| Carlo Descovich | Delegato del Direttore Sanitario di AUSL<br>di Bologna | AUSL di Bologna | Р |
| Danilo Di Diodoro * | Clinico specialista in psichiatria | in quiescenza | Р |
| Giuseppe Di Pasquale | Clinico specialista in cardiologia | Libero professionista | P |
| Carla Faralli | Esperto di bioetica | Università degli Studi di<br>Bologna | A |
| Carlo Feo | Delegato del Direttore Sanitario di AUSL<br>di Ferrara | AUSL di Ferrara | A |
| Maria Elena Flacco | Biostatistico | Università degli Studi di<br>Ferrara | P |
| Daniele Gallo * | Ingegnere clinico | AUSL di Reggio Emilia<br>IRCCS | P |

Allegato: elenco dei componenti del Comitato Etico presenti al momento dell'espressione del presente parere

**NOTA:** per qualsiasi successiva comunicazione relativa allo studio in oggetto è indispensabile fare riferimento al codice interno CE che identifica lo studio (indicato nell'oggetto) e alla data della seduta di valutazione.



### Comitato Etico di Area Vasta Emilia Centro

Il Comitato Etico di Area Vasta Emilia Centro della Regione Emilia-Romagna (CE-AVEC) è stato istituito presso IRCCS Azienda Ospedaliero—Universitaria di Bologna, Policlinico S.Orsola-Malpighi con delibera n. 6 del 10/1/2018. Il CE-AVEC opera in conformità al DM 12/05/2006 e al DM 08/02/2013.

| Filippo Giovanardi * | Clinico specialista in oncologia | AUSL di Reggio Emilia<br>IRCCS | Α |
|---|---|---|---|
| Marcello Govoni | Clinico specialista in reumatologia | AOU di Ferrara/Università<br>degli Studi di Ferrara | Α |
| Carlo Impallomeni | Delegato Direttore Sanitario AUSL Imola | AUSL di Imola | A |
| Maria Paola Landini | Direttore Scientifico dell'Istituto<br>Ortopedico Rizzoli | Istituto Ortopedico Rizzoli di<br>Bologna | A |
| Raffaele Lodi | Direttore Scientifico di IRCCS Istituto<br>delle Scienze Neurologiche<br>IRCCS-ISNB | IRCCS-ISNB Istituto delle<br>Scienze Neurologiche di<br>Bologna | Α |
| Susanna Maltoni | Esperto in dispositivi medici | IRCCS AOU di Bologna | Р |
| Renato Mantovani * | Esperto in materia assicurativa | Avvocato libero professionista | P |
| Gainluca Mazza* | Esperto in materia giuridica | IRST IRCCS di Meldola | Р |
| Monica Minardi * | Medico di medicina generale territoriale | MMG in convenzione con<br>AUSL Imola | P |
| Maria Cristina Morelli | Clinico specialista in gastroenterologia | IRCCS AOU di Bologna | Р |
| Danilo Orlandini * | Esperto in nutrizione | Libero professionista | P |
| Ilaria Panzini | Biostatistico | AUSL di Ferrara | Α |
| Angelina Passaro | Delegato del Direttore Sanitario di AOU<br>di Ferrara | AOU di Ferrara | Р |
| Michela Pastore * | Medico di medicina generale territoriale | MMG in convenzione con<br>AUSL Ferrara | P |
| Carla Pelusi | Clinico specialista in endocrinologia | IRCCS AOU di<br>Bologna/Università degli<br>Studi di Bologna | Р |
| Gian Matteo Rigolin | Clinico specialista in ematologia | AOU di Ferrara/Università<br>degli Studi di Ferrara | Р |
| Cesare Rossi | Esperto in genetica | IRCCS AOU di Bologna | Р |
| Fabrizio Sandri | Pediatra | AUSL di Bologna | Р |
| Luigia Scudeller | Delegato del Direttore Sanitario IRCSS<br>AOU di Bologna | IRCCS AOU di Bologna | Α |
| Savino Spadaro | Clinico specialista in anestesia-<br>rianimazione | AOU di Ferrara/Università<br>degli Studi di Ferrara | Р |
| Stefano Volpato | Clinico specialista in medicina interna/geriatria | AOU di Ferrara/Università<br>degli Studi di Ferrara | Р |

Allegato: elenco dei componenti del Comitato Etico presenti al momento dell'espressione del presente parere

**NOTA:** per qualsiasi successiva comunicazione relativa allo studio in oggetto è indispensabile fare riferimento al codice interno CE che identifica lo studio (indicato nell'oggetto) e alla data della seduta di valutazione.



### Comitato Etico di Area Vasta Emilia Centro

Il Comitato Etico di Area Vasta Emilia Centro della Regione Emilia-Romagna (CE-AVEC) è stato istituito presso IRCCS Azienda Ospedaliero-Universitaria di Bologna, Policlinico S.Orsola-Malpighi con delibera n. 6 del 10/1/2018. Il CE-AVEC opera in conformità al DM 12/05/2006 e al DM 08/02/2013.

| Claudio Zamagni | Clinico specialista in oncologia | IRCCS AOU di Bologna | A |
|---|---|---|---|
| Anita Zeneli * | Rappresentante dell'area delle professioni sanitarie interessata alla sperimentazione | IRST IRCCS di Meldola | P |

<sup>\*</sup> membri esterni

### Partecipano alla seduta i seguenti rappresentanti delle Segreterie (senza diritto di voto):

- Stefania Proni, Giacomo Chiabrando, Giovanni Comandini, Alessandra Brunetti, Elisabetta Chiodi, Urbano Briganti: Segreteria centrale presso IRCCS-Azienda Ospedaliero Universitaria di Bologna;
- Corrado Iacono, Paolo Dessi: Segreteria locale presso Azienda USL di Bologna;
- Renata Mesirca: Segreteria locale presso Azienda USL di Imola;
- Simonetta Gamberini, Daniele Righi, Rosa Celozzi: Segreteria locale presso Istituto Ortopedico Rizzoli;
- Marco Voci, Sandra Bombardi: Segreteria locale presso Azienda Ospedaliero Universitaria di Ferrara

Allegato: elenco dei componenti del Comitato Etico presenti al momento dell'espressione del presente parere

**NOTA:** per qualsiasi successiva comunicazione relativa allo studio in oggetto è indispensabile fare riferimento al codice interno CE che identifica lo studio (indicato nell'oggetto) e alla data della seduta di valutazione.



**DIREZIONE GENERALE** 

Al Prof. Carlo feo Direttore U.O. Chirurgia Provinciale AUSL Ferrara

E p.c

Alla Dott.ssa Ilaria Panzini Direttrice U.O. Qualità Accreditamento Ricerca Organizzativa

OGGETTO: Nulla osta e autorizzazione relativi allo studio osservazione con farmaco "L'efficacia della colangiografia fluorescente (NIRF-C) durante colecistectomia videolaparoscopica in urgenza nei pazienti affetti da colecistite acuta e nelle colecistectomie difficili (Colecistiti Acute)". PI Prof. Carlo Feo.

## Con riferimento allo studio in oggetto:

- richiamata la Delibera del Direttore Generale dell'Azienda USL di Ferrara n. 147 del 24/8/2018 di presa d'atto del riordino dei Comitati Etici della Regione Emilia Romagna e dell'istituzione del Comitato Etico indipendente dell'Area Vasta Emilia Centro;
- vista la valutazione positiva espressa in data 30/11/2021 da parte dell'U.O. Assistenza Farmaceutica Ospedaliera e Territoriale AUSL Ferrara dell'Azienda USL di Ferrara;
- preso atto che il Comitato Etico AVEC, con decisione assunta nella seduta telematica del 16/12 /2021, ha espresso parere favorevole alla conduzione dello studio a condizione che venisse dato riscontro alle richieste relative all'informativa privacy riportate nel verbale della seduta di cui sopra;
- preso atto che in data 11/01/2021 è stata inviata tramite email al Comitato Etico AVEC dallo Sperimentatore Principale dello studio, la documentazione richiesta di cui sopra;

rilevato che il Comitato Etico AVEC, a seguito della disamina della documentazione ricevuta, ha comunicato tramite email del 12/01/2022 a questa Azienda, di aver sciolto le riserve al parere

rilasciato in data 16/12/2021 di cui sopra;

considerato che in data 21/01/2022 si è provveduto da parte dell'UO Qualità, Accreditamento,

Ricerca Organizzativa ad inviare ad AIFA il protocollo e il modulo Moduli relativo al Registro degli

Studi Osservazionali (RSO);

considerato che, come dichiarato nel Modulo regionale Informazioni per la valutazione locale dello

studio e relative autodichiarazioni, firmato dal PI in data 06/11/2021, non sussistono spese

aggiuntive a carico dell'Azienda USL di Ferrara;

dato atto che lo studio no profit si configura come uno studio osservazionale con farmaco promosso

dall'Azienda USL di Ferrara e che sarà condotto presso l'UO Chirurgia Provinciale dell'Azienda USL

di Ferrara sotto la responsabilità del Prof. Carlo Feo in qualità di sperimentatore principale;

NULLA OSTA all'avvio delle attività dello studio in oggetto.

Contestualmente SI AUTORIZZA lo studio in oggetto:

individuando il Prof. Carlo Feo quale Sperimentatore principale nella conduzione dello studio presso

l'Azienda USL di Ferrara:

dando atto che lo studio non prevede emolumenti a favore dello sperimentatore e non emergono

costi ingiustificati derivanti dallo stesso posti in capo all'Azienda USL di Ferrara.

Firmato digitalmente da:

Monica Calamai

Responsabile procedimento: Luca Santini